CLINICAL TRIAL: NCT03008291
Title: His Bundle Pacing in Bradycardia and Heart Failure
Status: Recruiting | Type: Observational
Sponsor: Yong-Mei Cha (Other)
Responsible Party: Sponsor-Investigator, Yong-Mei Cha, M.D., Professor of Medicine, Mayo Clinic
Organization: Mayo Clinic (Other)
Other Study IDs: 16-005100
Record Dates: First submitted 2016-11-02; First posted 2017-01-02 (Estimated); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Bradycardia; Heart Failure
MeSH Terms: conditions — Bradycardia; Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Heart Failure Group: Patients who have any QRS duration and left ventricular ejection fraction (LVEF) ≤ 50% will be enrolled in this arm. The primary care physician will have recommended either PM, CRT-D Implantation, CRT-P Implantation, HIBP or LBAP (including HIBP/LBAP for patients with HF, for patients who have failed CRT implant or patients who are CRT non-responders) . (This is Standard of Care for this patient population; the procedures will occur even if the patient does not participate in the study.)
  Interventions: Procedure: CRT-D Implantation; Procedure: CRT-P Implantation
- Atrioventricular Block/Bradycardia Group: Patients who have developed second or third degree atrioventricular block (AV block) or bradycardia will be enrolled in this arm. The primary care physician will have recommended dual chamber pacemaker implantation. (This is Standard of Care for this patient population; the procedures will occur even if the patient does not participate in the study.)
  Interventions: Procedure: Dual Chamber Pacemaker Implantation

INTERVENTIONS:
Procedure: CRT-D Implantation — Cardiac resynchronization therapy defibrillator
  Groups: Heart Failure Group
Procedure: CRT-P Implantation — Cardiac resynchronization therapy pacemaker
  Groups: Heart Failure Group
Procedure: Dual Chamber Pacemaker Implantation
  Groups: Atrioventricular Block/Bradycardia Group

SUMMARY:
Participants in this study will either have heart failure (HF) and are scheduled to undergo pace maker (PM) implantation, cardiac resynchronization therapy pacemaker (CRT-P), cardiac resynchronization therapy defibrillator (CRT-D) implantation, His bundle pacing (HIBP) or left bundle area pacing (LBAP) (including HIBP/LBAP for patients with HF, for patients who have failed CRT implant or patients who are CRT non-responders), or have atrioventricular (AV) block or bradycardia and are scheduled to undergo dual chamber pacemaker implantation. In this study additional heart rhythm measurements will be collected during the implant procedure to better understand how His bundle and/or parahisian pacing (HISP) effects electrical conduction in the hearts of patients with HF or AV block.

The hypothesis is that His bundle or parahisian pacing (HISP) and left bundle area pacing (LBAP) may normalize atrioventricular (AV) conduction with a narrow combination of the Q wave, R wave and S wave (QRS complex) in functional bundle branch block or conduction delay in patients with heart failure (HF).

ELIGIBILITY:
Inclusion Criteria:

HF Group

* Clinically recommended to undergo PM, CRT-P, or CRT-D implantation or HIBP/LBAP (including HIBP/LBAP for patients with HF, for patients who have failed CRT implant or patients who are CRT non-responders)
* Any QRS duration
* LVEF ≤ 50%

AV Block/Bradycardia Group

* Recommended to undergo dual chamber pacemaker implantation
* Any AV block or Sinus Bradycardia

Exclusion Criteria:

* Age < 18 years
* Pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects will be recruited from the heart clinic at Mayo Clinic in Rochester, Minnesota.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2016-10; Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
QRS duration as measured by 12-lead ECG | Baseline to 6 months
  The normal duration (interval) of the QRS complex is 0.08 and 0.10 seconds (80 and 100 ms). When the duration is between 0.10 and 0.12 seconds it is intermediate or slightly prolonged. A QRS duration of greater than 0.12 seconds is considered abnormal.
QRS morphology as measured by 12-lead ECG | Baseline to 6 months
  Normal QRS width is 70-100 ms (a duration of 110 ms is sometimes observed in healthy subjects). The QRS width is useful in determining the origin of each QRS complex (e.g. sinus, atrial, junctional or ventricular).

CONTACTS AND LOCATIONS:
Overall Officials: Yong-Mei Cha, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No